CLINICAL TRIAL: NCT04185389
Title: Evaluation of CIN2+ Rates up to 120 Months After 48-Month Co-Testing (Long Term Follow up of HPV FOCAL Participants)
Brief Title: Long-Term Follow-Up of HPV FOCAL Participants
Acronym: HPV FOCAL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Cancer Agency (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Gina Ogilvie, Professor, University of British Columbia
Other Study IDs: H19-01584; 5R01CA221918-02 (NIH)
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Cervical Cancer
Keywords: hpv testing; cytology; human papillomavirus; cervix screening
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Control: Women in the original HPV FOCAL control arm who completed the 48 month exit screen (HPV/LBC co-test) and who had no CIN2+ detected during the trial or at trial exit will be invited to submit another LBC sample for HPV and cytology co-testing.
  Interventions: Other: HPV and cytology co-testing (via Liquid based collection device)

INTERVENTIONS:
Other: HPV and cytology co-testing (via Liquid based collection device) — Liquid-based cytology co-testing is a procedure in which that a cervical sample is taken, and can be co-tested for HPV and standard cytology at the same time. It is collected in the same way that a traditional Pap is collected

SUMMARY:
This FOCAL follow-up study aims to assess the long-term effectiveness and safety of primary HPV testing for cervical cancer screening. A cohort of participants from the original FOCAL study will be asked to see their health care provider to submit another cervical sample for cytology and HPV testing. This will permit evaluation of long term safety and effectiveness of primary HPV testing up to ten years after a participant's first screening in the FOCAL study and comparison of primary HPV testing to HPV and cytology co-testing.

DETAILED DESCRIPTION:
This study will evaluate the long-term effectiveness of primary HPV screening, with and without cytology co-testing at various time points and inform optimal algorithms for HPV-based cervical cancer screening. Specifically the project will compare rates of CIN2+ after primary HPV testing to rates of CIN2+ after baseline LBC testing followed by HPV and LBC "co-testing" at 48 months. We hypothesize that women who have a negative HPV result at baseline will have fewer CIN2+ lesions detected at 96 months or 120 months (or greater) after baseline than women who have a negative cytology (LBC) result at baseline, and who receive HPV/LBC co-testing at 48 months and at 96 months or greater after baseline.

Objectives

1. Determine detection rates of CIN2+ at approximately 48 months or 72 months (one sample only, depending on when women exited the trial) after the FOCAL 48 month exit HPV/LBC co-test screen in control arm women.
2. Compare CIN2+ rates from women in the intervention arm (HPV testing) at 48 month FOCAL HPV/LBC co-test screen, to CIN2+ rates of women in the control arm (LBC testing) receiving HPV/LBC co-testing up to 120 months or greater (if applicable). If CIN2+ outcomes are available beyond 120 months where available, this will be captured to ensure important endpoints are not missed because of a 120 month cut off. (For the remainder of this proposal, when indicating 120 months, this will include those with CIN2+ outcomes beyond 120 months).
3. Using passive follow-up by anonymized data linkage with the BC Cancer cervix screening registry, determine long term protection against CIN2+ up to 120 months after a negative HPV baseline result.

Women in the control arm (LBC testing at baseline) who completed the 48 month exit screen (HPV/LBC co-test) and who had no CIN2+ detected during the trial or at trial exit will be invited to participate. When women consented to participate in the HPV FOCAL trial, they were asked if they were interested in being contacted in the future for potential research studies related to cervical cancer. Women who indicated they would be interested and those who did not specifically state they did not want to be contacted, will be contacted.

An information letter will be sent to eligible participants with information describing the study. This information package will also include a link to a REDCap eConsent that has an eligibility survey and consent form. Interested women will be asked to complete this online eConsent form to give consent to participate. It is not possible to have face to face interactions with participants, given the nature of this trial, and electronic consent is the most feasible approach for this project. Electronic consent procedures will be followed per UBC guidelines and per US OHRP "Use of Electronic Consent" guidelines. https://www.fda.gov/media/116850/download.

After eligibility has been confirmed, women will be directed to their usual HCP for a cervical sample collection with Liquid based cytology, permitting for both HPV and cytology testing on the same sample.

All LBC samples will be sent to the PHL for HPV and cytology testing.

In order to compare the results of post- 48month trial exit follow-up for women in the FOCAL control arm (who had baseline LBC testing) to women in the FOCAL intervention arm (who had baseline HPV testing), a data linkage will be conducted between the FOCAL study database, the Cervix Screening Program Registry and the BC Cancer Registry, using BC Cancer Registry Data Linkage established procedures.

ELIGIBILITY:
Inclusion Criteria:

* Previous HPV FOCAL study, control arm participants who completed 48 month FOCAL LBC/HPV co-testing with no CIN2+ detected at trial exit
* Resident of BC
* <69 years of age (upper age limit for routine screening per BC Cancer Cervix Screening program)
* No history of CIN2+ since FOCAL study exit or in the last 5 years
* Has not had a hysterectomy
* Has never had a diagnosis of invasive cervical cancer

Ages: 30 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists entirely of participants from a previous RCT.
Sampling Method: Non-Probability Sample
Enrollment: 1710 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of CIN2+ | 120 months
  Moderately abnormal cells are found on the surface of the cervix

CONTACTS AND LOCATIONS:
Overall Officials: Gina Ogilvie, MD, MSc FCFP DrPH, Principal Investigator — University of British Columbia; Laurie Smith, MPH, Study Director — BC Cancer
Locations (1):
- Women's Health Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No